(General Organization) - Jeddah

#### Title of Research:

A Randomized Controlled Trial Comparing Blood Glucose Control Intraoperative Between Insulin Drip vs. Insulin **Boluses** 

#### A. Purpose of the Research:

The primary objective is to compare blood glucose control intraoperatively between patients who receive insulin drip and patients who receive insulin boluses during adult cardiac surgery. The secondary objective is to evaluate the incidence of hypoglycemic events and the need for insulin adjustments during surgery.

#### B. Description of the Research:

Adult patients (age  $\geq$  18 years) undergoing cardiac surgery with preoperative blood glucose levels between 80-180 mg/dL. A total of 200 adult patients will be randomly assigned to each arm. Patient will be randomized to either group A (Insulin drip will be administered at a starting rate of 2 units/hour and titrated to maintain blood glucose levels between 80-180 mg/dL), or group B (Insulin boluses will be administered every 30 minutes to maintain blood glucose levels between 80-180 mg/dL). The overall study duration is estimated to be 4 years.

#### C. Potential Benefits:

This randomized controlled trial will provide valuable information on the optimal method for achieving blood glucose control intraoperatively. The results of this study may help improve patient outcomes and reduce the incidence of postoperative complications.

# D. Potential Risks and Discomforts:

Both methods of insulin delivery are already in use and FDA approved. The possible adverse reaction include hypglycemia, allergic reaction, and extravasation at injection site

### E. Voluntary Participation:

Participation in this study is voluntary. You will not suffer penalty nor loss of any benefits to which you are entitled for, if you decide not to participate.

Significant new findings developed during the course of the study, which might be expected to affect your willingness to continue to participate in the study, will be provided to you. A signed copy of consent form

#### عنوان البحث:

دراسة عشوائية بهدف تقييم مستوى السكر في الدم باستخدام جرعات الانسولين المتفرقة مقارنة بجرعات الانسولين المتواصلة . المتواصلة أ. الغرض من البحث:

مقارنة مستوى السكر في الدم بعد اعطاء الانسولين بطريقتين مختلفه خلال عمليات جراحة القلب المفتوح

### ب. وصف البحث:

تستهدف الدراسة المرضى البالغين اكبر من ١٨ عام والذين يبلغ مستوى السكر في الدم لديهم من ٨٠ – ١٨٠ مج/دل لاضافتهم الى احد المجموعتين العلاجية. الاولى يتم استخدام جرعات الانسولين المتواصلة مع قياس مستوى السكر كل نصف ساعة وستكون مدة الدراسة تقريبا ٤ سنوات

# ج الفوائد المحتملة:

تهدف هذة الدراسة الى اعطاء معلومات مهمة عن الطريقة الأمثل للتحكم في مستوى سكر الدم أثناء العملية الجراحية و ذلك قد يحسن من نتائج المرضى مما قد يؤدي الي تقليل للمضاعفات المتوقعة

# د. المخاطر والانزعاجات المحتملة:

الطريقتين مستخدمة في العلاج ومرخصة من هيئة الغذاء والدواء. والمضاعفات المحتملة تشمل هبوط في مستوى السكر في الدم، رد فعل تحسسي، تجمع دموي في مكان الحقن

# ه. المشاركة الطوعية:

المشاركة في هذه الدراسة طوعية وإذا قررت عدم المشاركة فإنك لن تتعرض لأية مضايقات أو لفقدان حقك المشروع في

سيتم إبلاغك بأية نتائج جديدة هامة تظهر خلال سير الدراسة والتي قد تؤثر في رغبتك في الاستمرار بالمشاركة في هذه الدر اسة سيتم تز و يدك بنسخة مو قعة من هذا الإقر ار

This Informed Consent Form (ICF) is approved by the Institutional Review Board at ICF Version No.: 2.0 Date: 16-10-2023

IRB #.: 2023-45

The Informed Consent Approved By IRB

From: 04 November 2024 To: 04 November 2025 Approval Date:

(General Organization) - Jeddah

will be given to you.

# F. Alternative to Participation and Withdrawal (if applicable):

Withdrawal from or not participating in this research study will not affect your ability to obtain alternative methods of medical care available at King Faisal and Research Centre (General Organization) - Jeddah

#### G. Confidentiality:

Your identity and medical record, as a participant in this research study, will remain confidential with respect to any publications of the results of this study. However, your medical record may be reviewed by the principal investigator/ delegate involved in this research, the Institutional Review Board, or the agency sponsoring this research in accordance with applicable laws and regulations.

#### H. Compensation:

In the event of injury resulting from participation in this research study, KFSH&RC-J will make available to you, including admission, if required, its hospital facilities and professional attention. Financial compensation from KFSH&RC-J, however, is not available.

#### I. Reimbursements:

KFSH&RC-J will not reimburse the participant for participation in the study.

#### J. Contact Person(s):

For any specific questions regarding this study or in the event of a research-related injury, please contact the pricipal investigator/delegate, <u>Dr Mohammed</u> Alrefai

telephone No. 012667-7777 Ext. 49796

For general questions concerning research at

# و. البدائل عن المشاركة والانسحاب من المشاركة (إن وجد):

إن قرارك بعدم الإشتراك أو بالانسحاب من الدراسة لن يؤثر على تاقيك لخدمات علاجية بديلة متوفرة في مستشفى الملك فيصل التخصصي و مركز الابحاث بجدة (مؤسسة عامة).

# ز. السرية:

كمشارك في هذه الدراسة ستكون هويتك ومحتويات ملفك الطبّي سرية في جميع المنشورات المتعلقة بنتائج الدراسة. إلا إنه يمكن لكل من الباحث الرئيسي/نائبه،أو المجلس التقييمي للأبحاث،أو الجهة الداعمة للدراسة الاطلاع على ملفك الطبي و ذلك في حدود النظم والقوانين المطبقة بهذا الخصوص.

# ح التعويضات:

في حالة حدوث أي ضرر لا قدر الله من جراء مشاركتك بهذه الدراسة؛ سيتكفل مستشفى الملك فيصل التخصصي ومركز الأبحاث بجدة بتقديم العناية الطبية اللازمة أو التنويم في المستشفى إن لزم الأمر، ولكنه لا يوجد أي تعويضات مالية.

### ط التعويض المالى:

لا يلتزم مستشفى الملك فيصل التخصصى و مركز الأبحاث بجدة (مؤسسة عامة) بدفع أى تعويض مالي مقابل المشاركة في البحث.

# ي. الأشخاص الذين يمكن الاتصال بهم:

للأسئلة العامة المتعلقة بالبحوث بمستشفى الملك فيصل التخصيصي ومركز الأبحاث بجدة يرجى الإتصال على منسقة

•••••

This Informed Consent Form (ICF) is approved by the Institutional Review Board at

ICF Version No.: 2.0 Date: 16-10-2023

IRB #.: 2023-45

The Informed Consent Approved By IRB

From: 04 November 2024 To: 04 November 2025

(General Organization) - Jeddah

KFSH&RC-Jeddah, you may call the research coordinator telephone # 012667-7777 Ext. 43872 or the Institutional Review Board telephone #012667-7777 Ext. 62984.

الأبحاث على هاتف رقم ١٢٦٦٢٧٧٧٧ تحويلة رقم ٤٣٨٧٢ أو الاتصال على رئيس مجلس تقييم الابحاث/نائبه على هاتف رقم ٦٢٩٨٤.

K. I, the principal investigator/delegate

confirm that I have fully explained to the above patient's gaurdian the nature and purpose of the foregoing study, possible alternative methods of treatment, the benefits reasonably to be expected, the attendant discomforts and risks involved, the possibility that complications may arise as a result thereof.

It is my understanding that the above patient's gaurdian understands the nature, purposes, benefits, and risks of participation in this research before signing of this informed consent. I have also fully and completely answered all questions the above patient's gaurdian has with respect to such research.

ك. أقر أنا الباحث الرئيسي/نائبه

بأنني قد شرحت بصورة كاملة للمريض /ولي أمرة طبيعة الدراسة, والغرض منها, والطرق العلاجية البديلة ، والفوائد المحتملة, والمخاطر والانزعاجات المتوقعة ، والمضاعفات التي قد تحدث كنتيجة للدراسة.

من المفهوم لديّ بأن المريض المذكور أعلاه /ولي أمره قد فهم طبيعة الدراسة والهدف منها والفوائد والمخاطر المترتبة على المشاركة فيها قبل توقيعه على الموافقة بالمشاركة.

وقد قمت بالإجابة على جميع أسئلة المريض *إو*لي أمره إجابة واضحة ومرضية.

Human Subject Acknowledgment to participate in Research

إقرار المشارك بالموافقة على المشاركة بالبحث

This Informed Consent Form (ICF) is approved by the Institutional Review Board at

ICF Version No.: 2.0 Date: 16-10-2023

IRB #.: 2023-45

The Informed Consent
Approved By IRB

From: 04 November 2024 To: 04 November 2025

Approval Date:

(General Organization) - Jeddah

L. I, the the participate acknowledge that I have read (or it had been explained to me in a clear language) the attached Research Participant Information Form and

has explained to me the nature and purpose of this study in this form, as well as any reasonably expected benefits, possible alternative methods of treatment, the attendant discomforts and risks reasonably expected, and the possibility that complications from both known and unknown causes may arise as a result thereof. I have had the opportunity to ask any questions I had regarding this study and all those questions were answered to my satisfaction. I also agree that blood, body fluids/tissues, and fetus tissues may be sampled for research analyses and related purposes. I am unaware of any preexisting medical or emotional problem which would make it unwise for me to participate in this research.

Based on the above mentioned information I voluntarily accept participation in this research study and I understand that I am free to withdraw this consent and discontinue my participation in this study at any time. The consequences and risks, if any, which might be involved if I decided to discontinue my participation have been explained to me. I understand that such withdrawal will not affect my ability to receive any medical care to which I might be otherwise entitled.

ل. أقر أنا المشارك بأنني قد قرأت (أو قد شُرحت لي بلغة واضحة) جميع المعلومات الموجودة في نموذج الإقرار بالموافقة على المشاركة بالأبحاث وإن

قد أوضح لي ماهية الدراسة في هذا النموذج, والغرض منها, والفوائد المرجوة منها, والطرق العلاجية البديلة لها, والمخاطر أوالانز عاجات المتوقع حدوثها, وكذلك احتمال حدوث مضاعفات لأسباب معروفة أو غير معروفة نتيجة لذلك. كما أنه قد أتيحت لي الفرصة الكافية لطرح أي سؤال يتعلق بالدراسة وتلقيت الإجابات الكافية. كما أوافق على أنه قد تؤخذ عينات من الدم, سوائل أو أنسجة الجسم, أو أنسجة من الجنين وذلك لأغراض تحليلية ومتعلقة بالدحث.

كما أقر بأنني لا أعاني من أي مشاكل طبية أو نفسية معروفة لدي بحيث قد يكون من غير الحكمة أن أشارك بهذه الدراسة.

بناء على ما سبق وبمحض إرادتي فإني أتطوع بالمشاركة في هذه الدراسة, وأفهم أن لي مطلق الحرية بسحب موافقتي وقطع مشاركتي بالدراسة في أي وقت. هذا وقد شرحت لي جميع العواقب والمخاطر المترتبة (إن وجدت) عن انسحابي من الدراسة. كما أفهم بأن انسحابي من هذه الدراسة لن يؤثر في حقي في تلقّى العناية الطبية اللازمة التي أستحقها في الأحوال العادية.

#### Title of Research:

A Randomized Controlled Trial Comparing Blood Glucose Control Intraoperative Between Insulin Drip vs. Insulin Boluses عنوان البحث : دراسة عشمائرا

دراسة عشوانية بهدف تقييم مستوى السكر في الدم باستخدام جرعات الانسولين المتفرقة مقارنة بجرعات الانسولين المتواصلة

This Informed Consent Form (ICF) is approved by the Institutional Review Board at

ICF Version No.: 2.0 Date: 16-10-2023

IRB #.: 2023-45

The Informed Consent
Approved By IRB

Approval Date: From: 04 November 2024 To: 04 November 2025

| Patient's | Addressograph |
|-----------|---------------|

(General Organization) - Jeddah

| (General Organization) - Jeddan | |
|---|---|
| Name of Participant: | اسم المشارك: |
| Name of individual signing the consent form: | اسم الموقع على هذا الإقرار: |
| Gaurdian's Relation: | صفة ولي الأمر: |
| Signature: | التوقيع: |
| Date: | التاريخ: |
| Witness Name: | اسم الشاهد : |
| Signature/(National I.D./Iqama/Hospital I.D. No.): | التوقيع/ (رقم الهوية/ الإقامة/ الرقم الوظيفي): |
| Date / Time: | التاريخ/ الوقت: |
| Signature of Principal Investigator/ Delegate | توقيع الباحث الرئيسي/نائبه |
| Name: | וצו וואים: |
| I.D. No.: | الرقم الوظيفي: |
| Title: | الوظيفة: |
| Date: | التاريخ: |

| This Informed Consent Form (ICF) is | ICF Version No.: 2.0 | Date: 16-10-2023 |
|---|---|---|
| approved by the Institutional Review Board at | IRB #.: 2023-45 | The Informed Consent |

Approval Date: From: 04 November 2024 To: 04 November 2025

Approved By IRB